CLINICAL TRIAL: NCT04892992
Title: Dialogical Family Guidance in Families With a Child With Neurodevelopmental Disorders
Brief Title: Dialogical Family Guidance for Neurodevelopmental Disorders
Acronym: DFG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diana Cavonius-Rintahaka (Other)
Responsible Party: Sponsor-Investigator, Diana Cavonius-Rintahaka, PhD candidate, Tampere University
Organization: Tampere University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106/13/03/03/2012
Record Dates: First submitted 2021-05-07; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Family Dynamics
Keywords: Dialogical family guidance; family health; neurodevelopmental disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Intervention group I were delivered DFG immediately and Intervention group II were delivered DFG after three months.
Who Masked: Participant
Masking Description: Intervention group I were delivered DFG immediately, and Intervention group II were delivered DFG after three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group I (Experimental): 6 sessions of intervention DFG starting at once (baseline). After DFG treatment as usual at Helsinki University hospital. The change between before the intervention (baseline) and after the intervention (3 months later) is being assessed.
  Interventions: Behavioral: DFG
- Intervention group II (Experimental): 6 sessions of intervention DFG starting 3 months after baseline (3 months on waiting list). Between baseline and 3 months waiting list families were getting treatment as usual at Helsinki University hospital. The change between baseline - after 3 months waiting list (3 months from baseline)/ before the intervention - and after intervention (6 months from baseline) is being assessed. Also the difference between Intervention group I and II is assessed.
  Interventions: Behavioral: DFG

INTERVENTIONS:
Behavioral: DFG

SUMMARY:
Previous studies have highlighted the need to offer targeted effective interventions to strengthen the wellbeing of all family members in families with children with neurodevelopmental disorders (NDD). Interventions for this target group requires development and research. A new family intervention, Dialogical Family Guidance (DFG) was tested in this study. All families received DFG intervention ( 6 meetings ).

DETAILED DESCRIPTION:
Previous studies have highlighted the need to offer targeted effective interventions to strengthen the wellbeing of all family members in families with children with neurodevelopmental disorders (NDD). Interventions for this target group requires development and research. A new family intervention, Dialogical Family Guidance (DFG) was tested in this study.

Fifty families of children with NDD were randomized into two intervention groups. Intervention group I were delivered DFG immediately, and Intervention group II were delivered DFG after three months. Family functionality, health and support (FAFHES), SDQ and the 5-15-questionnaire and DFG parent questionnaires were used to collect data at baseline, after three and six months. Fifty families were invited to the study. Thirty-four families completed the study. A comparison were made between Intervention group I and II.

ELIGIBILITY:
Inclusion Criteria:

* clinical neurodevelopmental disorder diagnosis (eg ADHD, ASD, tics, language disorders)
* the child is aged between 4-16 years
* parent have adequate Finnish language skills
* parents are biological parents or step-parents of the child

Exclusion Criteria:

* the child is under 4 or over 16 years old
* parents do not have adequate Finnish language skills

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The Family Function, Health and Social Support - scale (FAFHES) | Baseline measure before DFG family intervention starts
  The FAFHES questionnaire contains three sections; family functionality (19 items), family health (23 items), and family support provided by professionals (21 items). All the items are measured on a Likert scale ranging from 1-6 (I disagree totally, I disagree, I disagree somewhat, I agree somewhat, I agree, I agree totally). Family functionality, family health and family support were seen as poor if the median was 1.00-2.7, moderate if it was 2.8-4.5, and good if it was 4.6-6.0.45. Parent questionnaire. 1=I totally disagree.....6=I absolutely agree. Higher scores mean worse outcome.
The Family Function, Health and Social Support Scale (FAFHES) | 3 months after baseline measure, when intervention is finished. Change is being assessed.
  The FAFHES questionnaire contains three sections; family functionality (19 items), family health (23 items), and family support provided by professionals (21 items). All the items are measured on a Likert scale ranging from 1-6 (I disagree totally, I disagree, I disagree somewhat, I agree somewhat, I agree, I agree totally). Family functionality, family health and family support were seen as poor if the median was 1.00-2.7, moderate if it was 2.8-4.5, and good if it was 4.6-6.0.45. Parent questionnaire. 1=I totally disagree.....6=I absolutely agree. Higher scores mean worse outcome.
The Family Function, Health and Social Support Scale (FAFHES) | 6 months after baseline follow up. Change is being assessed.
  The FAFHES questionnaire contains three sections; family functionality (19 items), family health (23 items), and family support provided by professionals (21 items). All the items are measured on a Likert scale ranging from 1-6 (I disagree totally, I disagree, I disagree somewhat, I agree somewhat, I agree, I agree totally). Family functionality, family health and family support were seen as poor if the median was 1.00-2.7, moderate if it was 2.8-4.5, and good if it was 4.6-6.0.45. Parent questionnaire. 1=I totally disagree.....6=I absolutely agree. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
The Dialogical Family Guidance (DFG) - questionnaire | 3 months after baseline measure, when intervention is finished.
  The DFG-questionnaire was developed for this study to obtain information and parents' experiences about the DFG family intervention. The questionnaire include 14 items. Questions about the content and recommendation of DFG sessions were for example: "Did you get practical tips for daily life?" (1= yes absolutely….5=not at all) and "Would you recommend DFG to other parents?" (1=yes absolutely….4=no). The following semi-structured open-ended question was included in the DFG-questionnaire: Could you describe your experiences, comments or/and ideas about how to improve DFG? Parents filled the questionnaire after completing the DFG process (six meetings). Most questions were opinions about DFG, but when questions about "Did you get help from DFG?" 1=very much.... 5=not at all
The Strengths and Difficulties Questionnaire (SDQ) | Baseline measure before DFG family intervention starts
  SDQ measures the changes in child's behavior. 25 items with 3-point likert scale; Not true (0)- Somewhat true (1) - Certainly true (2). Parent questionnaire. Higher scores mean worse outcome considering the child with neurodevelopmental disorder.Highest scores 50 - lowest 0. Total score16-40 = high risk for abnormalities.
The Strengths and Difficulties Questionnaire (SDQ) | 3 months after baseline measure, when intervention is finished. Change is being assessed.
  SDQ measures the changes in child's behavior. 25 items with 3-point likert scale; Not true (0)- Somewhat true (1) - Certainly true (2). Parent questionnaire. Higher scores mean worse outcome considering the child with neurodevelopmental disorder.Highest scores 50 - lowest 0. Total score16-40 = high risk for abnormalities.
The Strengths and Difficulties Questionnaire (SDQ) | 6 months after baseline follow up. Change is being assessed.
  SDQ measures the changes in child's behavior. 25 items with 3-point likert scale; Not true (0)- Somewhat true (1) - Certainly true (2). Parent questionnaire. Higher scores mean worse outcome considering the child with neurodevelopmental disorder.Highest scores 50 - lowest 0. Total score16-40 = high risk for abnormalities.
Parent Questionnaire for Evaluation of Development and Behaviour in 5-15-year old Children, 5-15 (FTF, Five - to - Fifteen) | Baseline measure before DFG family intervention starts
  Parent Questionnaire for evaluation of development and behaviour in 5-15-year old children. 181 items. Three point likert scale; Not true (0) - Somewhat true (1)- Certainly true (2). Higher scores mean worse outcome considering the child. 0-13 scores normal and 17-40 scores mean abnormal result/abnormal
Parent Questionnaire for Evaluation of Development and Behaviour in 5-15-year old Children, 5-15 (FTF, Five - to - Fifteen) | 3 months after baseline measure, when intervention is finished. Change is being assessed.
  Parent Questionnaire for evaluation of development and behaviour in 5-15-year old children. 181 items. Three point likert scale; Not true (0) - Somewhat true (1)- Certainly true (2). Higher scores mean worse outcome considering the child. 0-13 scores normal and 17-40 scores mean abnormal result/abnormal
Parent Questionnaire for Evaluation of Development and Behaviour in 5-15-year old Children, 5-15 (FTF, Five - to - Fifteen) | 6 months after baseline follow up. Change is being assessed.
  Parent Questionnaire for evaluation of development and behaviour in 5-15-year old children. 181 items. Three point likert scale; Not true (0) - Somewhat true (1)- Certainly true (2). Higher scores mean worse outcome considering the child. 0-13 scores normal and 17-40 scores mean abnormal result/abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Diana Cavonius-Rintahaka, MhSc, Principal Investigator — Tampere University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cavonius-Rintahaka D, Roos M, Aho AL. The effectiveness of a dialogical family guidance intervention regarding child treatment response in families with a child with neurodevelopmental disorders. BMC Psychol. 2024 Apr 5;12(1):189. doi: 10.1186/s40359-024-01706-9. PMID 38580992